CLINICAL TRIAL: NCT05703581
Title: Application of "Heidelberg Triangle" Dissection in Pancreatoduodenectomy and Distal Pancreatectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: Huadong Hospital to Fudan
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pancreatoduodenectomy; Periampullary Carcinoma; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PD(TRIANGLE): Patients with pancreatic head cancer or periampullary cancer underwent "Heidelberg Triangle" dissection (TRIANGLE operation) combined with Pancreatoduodenectomy and standard lymphadenectomy
  Interventions: Procedure: TRIANGLE operation
- PD(non-TRIANGLE): Patients with pancreatic head cancer or periampullary cancer underwent pancreatoduodenectomy with standard lymphadenectomy
- DP(TRIANGLE): Patients with carcinoma of the body and tail of the pancreas underwent "Heidelberg Triangle" dissection (TRIANGLE operation) combined with distal pancreatectomy and standard lymphadenectomy
  Interventions: Procedure: TRIANGLE operation
- DP(non-TRIANGLE): Patients with carcinoma of the body and tail of the pancreas underwent distal pancreatectomy with standard lymphadenectomy

INTERVENTIONS:
Procedure: TRIANGLE operation — dissection the region composed of common hepatic artery (CHA), superior mesenteric artery (SMA) and superior mesenteric vein (SMV)
  Groups: DP(TRIANGLE); PD(TRIANGLE)

SUMMARY:
Aim of the study :

To evaluate the effect and safety of "Heidelberg Triangle" dissection (TRIANGLE operation) combined with Pancreatoduodenectomy or Distal Pancreatectomy on the prognosis of pancreatic cancer and periampullary cancer .

Methods :

Patients who underwent pancreatoduodenectomy or Distal Pancreatectomy between 01 September 2016 and 30 December 2022 will be included in this retrospective analysis. 3D reconstruction is performed with preoperative enhanced CT, then the region of "Heidelberg Triangle" is categorized . The operation is completed by the same operation team. According to the operation mode, patients were divided into TRIANGLE group and non-TRIANGLE group and And followed up until recurrence, death or missed.

DETAILED DESCRIPTION:
The "Heidelberg Triangle" is an anatomical area composed of Common hepatic artery (CHA), superior mesenteric artery (SMA) and superior mesenteric vein (SMV).

This area is considered to be the common site of recurrence after pancreatic surgery.

Recent studies have shown that TRIANGLE operation can improve the state of the cutting edge and has potential value in improving the prognosis. However, the data on recurrence and survival rate of pancreatic cancer and periampullary cancer after TRIANGLE operation are insufficient.

The aim of the present study is to evaluate the effect and safety of "Heidelberg Triangle" dissection combined with Pancreatoduodenectomy or Distal Pancreatectomy on the prognosis of pancreatic cancer and periampullary cancer .

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed by preoperative imaging and auxiliary examination as resectable or borderline resectable pancreatic malignant tumor or periampullary carcinoma who underwent pancreatoduodenectomy or distal pancreatectomy, with or without TRIANGLE operation.
2. Patients who have no serious abnormalities of blood system, heart and lung function and immune deficiency and can tolerate surgery.
3. Be able to comply with the research visit plan and other program requirements

Exclusion Criteria:

1. Patients accompanied by other systemic malignancies.
2. Central nervous system disease, mental disease, unstable angina pectoris, congestive heart failure, serious arrhythmia and other uncontrollable serious diseases, unable to tolerate surgery.
3. Pregnant and lactating women.
4. Any condition that may impair the safety of patients or the integrity of research data, including serious medical risk factors, medical conditions, and laboratory abnormalities.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed by preoperative imaging and auxiliary examination as resectable or borderline resectable pancreatic malignant tumor or periampullary carcinoma who underwent undergo pancreatoduodenectomy or distal pancreatectomy, with or without TRIANGLE operation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) | up to 72 months
  from the date of surgery to the first radiographic or pathologic evidence of recurrence.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 72 months
  from the date of diagnosis to death or last follow up
Surgical Morbidity | 90 postoperative days
  including postoperative pancreatic fistula (B/C), bile leakage (B/C), delayed gastric emptying (B/C), postpancreatectomy haemorrhage (B/C), postoperative chyle leak (B/C), postoperative intra-abdominal infection.

CONTACTS AND LOCATIONS:
Overall Officials: Chongyi Jiang, PhD, Principal Investigator — Huadong Hospital
Locations (1):
- Huadong Hospital affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No